CLINICAL TRIAL: NCT06352853
Title: A Comparative Study Between the Use of Scalpel Versus Diathermy in Opening the Transverse Abdominal Skin Incision During Cesarean Section
Brief Title: Scalpel Versus Diathermy in Transverse Abdominal Skin Incision During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mostafa Mohammed Refaay El shemy, Lecturer at Obstetrics and Gynecology department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Diathermy and skin incision cs
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Skin Wound
Keywords: Diathermy-Scalpel-skin incision-Cesarean section

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Scalpel Group (Active Comparator): A skin incision is made by traditional method, with proper homeostasis by application of pressure to skin blood vessels and by ligating the subcutaneous bleeding as well as using of diathermy on coagulation mode. Then,the scalpel was used to reach peritoneum.
  Interventions: Other: Skin incision in Cesarean Section by Scalpel
- Group 2: Diathermy Group (Active Comparator): A skin incision is made using a small flat blade pen electrode, set on cutting mode and delivering a 120-wat (maximum) sinusoidal current, electrosurgical cutting performed without pressure or mechanical displacement. Then, we used the scalpel to reach peritoneum.
  Interventions: Other: Skin incision in Cesarean Section by Diathermy

INTERVENTIONS:
Other: Skin incision in Cesarean Section by Diathermy — Skin incision by diathermy
  Arms: Group 2: Diathermy Group
Other: Skin incision in Cesarean Section by Scalpel — Skin incision by scalpel
  Arms: Group 1: Scalpel Group

SUMMARY:
This study aims to compare between using of diathermy versus scalpel in making skin incision during cesarean section to judge the variations in incisional time, incisional blood loss, postoperative pain, wound healing and wound complications.

DETAILED DESCRIPTION:
Surgical scalpels are traditionally used for skin incisions during a Caesarean delivery; the great evolutions in electrosurgical devices bring an alternative method for skin incision by the usage of cutting diathermy.

The current comparative study was conducted in Kasr Al-Ainy hospital obstetric theaters between January 2022 and June 2022. Consents were obtained from all participants. 120 participants were included in this study, divided into 2 groups 60 in each group;Diathermy group and scalpel group respectively .

• Randomization achieved using computer generated randomization sequences. Allocation was in 1:1 ratio

In both groups:

1. Pre-operative: patients received cefoperazone 1gm intravenous. In case of penicillin allergy, they received clindamycin intravenous.
2. A Pfannenstiel skin incision was made taken down through the subcutaneous tissue, rectus sheath and dissected from rectus muscle until peritoneum was visualized,

   * In scalpel group; an incision made by traditional method, with proper homeostasis by application of pressure to skin blood vessels and by ligating the subcutaneous bleeding as well as using of diathermy on coagulation mode. Then, the investigators used the scalpel to reach peritoneum.
   * In diathermy group; incision made using a small flat blade pen electrode, set on cutting mode and delivering a 120-wat (maximum) sinusoidal current, electrosurgical cutting performed without pressure or mechanical displacement. Then, the investigators used the scalpel to reach peritoneum.
   * The study compared incisional time by using digital clock, time established as follows: when skin incision made, the surgeon called out "start the clock". After opening the rectus sheath, the surgeon called out" stop the clock". Incision time is the difference between "start" and "stop".

   Also incision blood loss was calculated by weighing the swabs pre and postoperatively (1mg = 1ml). In incisional site no suction was used.

   •Also hemodynamic changes were compared between both groups that include: blood pressure (systolic blood pressure, diastolic blood pressure and mean arterial blood pressure), pulse, oxygen saturation and electrocardiogram (ECG) changes.
3. Intra-operative: patient received Diclofenac sodium 50-100 mg intramuscular and postoperatively, they received paracetamol vial /6 hours in both groups.

Closure of the skin in all cesarean sections was done by proline 2.0 for assessment of wound healing and complications.

Postoperatively, the postoperative pain was compared for 24 hours by visual analogue scale (VAS) score, It is 11 points numeric scale ranges from "0" representing one pain extreme (e.g.: no pain) to "10" representing the other pain extreme (e.g.: "pain as bad as you can imagine" or "worst pain imaginable") this will be recorded at 2,4, 6,8, 10,12, 24 hours postoperatively.

Lastly, wound healing was compared in both groups and complications like seroma, hematoma, ecchymosis, dehiscence and infection. The presence or absence of infection was assessed by Southampton grading system as following:

G0: normal wound healing, G1: normal healing with mild bruising or erythema, G2: erythema plus other signs of inflammation, G3: clear or serosanguinous discharge and G4: purulent discharge and in this case wound culture was performed.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean section.
* Women with body mass index less than 30.
* Transverse skin incision.

Exclusion Criteria:

* Women with medical disorder that can affect wound healing as diabetes, hypertension, chronic anemia and with chronic skin conditions as psoriasis and eczema.
* Women with Autoimmune disorders.
* Cardiac patients on pacemakers and patients on anticoagulants.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Skin incision time in scalpel versus diathermy group | 5 months
  The incision time was estimated by using digital clock, time established as follows: when skin incision made, the surgeon called out "start the clock". After opening the rectus sheath, the surgeon called out" stop the clock". Incision time is the difference between "start" and "stop".
Estimation of incision blood loss in both groups | 5 months
  incision blood loss volume was measured by weighing the swabs pre and postoperatively (1mg = 1ml).

SECONDARY OUTCOMES:
Postoperative pain in both groups | 5 months
  Evaluation of post operative pain for 24 hours by visual analogue scale
Postoperative wound healing in both groups | 5 months
  Postoperative wound complications like seroma, hematoma, ecchymosis, dehiscence (separation of the subcutaneous tissues with skin) and infection. The presence or absence of infection was assessed by Southampton grading system as following: G0: normal wound healing, G1: normal healing with mild bruising or erythema, G2: erythema plus other signs of inflammation, G3: clear or serosanguinous discharge and G4: purulent discharge and in this case wound culture was performed.

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa El Shemy, MD, Principal Investigator — Cairo University
Locations (1):
- Shaimaa El Shemy, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 10 years